CLINICAL TRIAL: NCT00118742
Title: A Randomized, Open-label Study of the Effect of a Long-term Calcineurin Inhibitor-free Maintenance Regimen With CellCept and Sirolimus on Preservation of Renal Function and Prevention of Acute Rejection in Recipients of an Orthotropic Liver Transplant
Brief Title: Liver Spare the Nephron (STN) Study - A Study of CellCept (Mycophenolate Mofetil) and Sirolimus in Recipients of a Liver Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18423
Record Dates: First submitted 2005-06-30; First posted 2005-07-12 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Tacrolimus; Cyclosporine; Sirolimus

ARMS (2):
- CellCept + CNI (tacrolimus or cyclosporine) (Experimental)
  Interventions: Drug: mycophenolate mofetil [CellCept]; Drug: Tacrolimus; Drug: Cyclosporine
- CellCept + sirolimus (Active Comparator)
  Interventions: Drug: mycophenolate mofetil [CellCept]; Drug: Sirolimus

INTERVENTIONS:
Drug: mycophenolate mofetil [CellCept] — 1-1.5 g orally or intravenously twice daily
Drug: Tacrolimus — As prescribed, for 12 months
  Arms: CellCept + CNI (tacrolimus or cyclosporine)
Drug: Cyclosporine — As prescribed, for 12 months
  Arms: CellCept + CNI (tacrolimus or cyclosporine)
Drug: Sirolimus — 2-4 mg orally once daily for 9-11 months
  Arms: CellCept + sirolimus

SUMMARY:
This two-arm study will assess the efficacy and safety of a long-term calcineurin inhibitor-free maintenance regimen with CellCept and sirolimus in recipients of an orthotropic liver transplant. Patients will be randomized to receive either CellCept 1-1.5 g twice daily (BID) + tacrolimus + cyclosporine, or CellCept 1-1.5 g BID + sirolimus. The anticipated time on study treatment is 1 to 2 years, and the target sample size is 100 to 500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-74 years of age
* Single primary liver transplant from a deceased donor
* CellCept plus tacrolimus or cyclosporine from time of transplantation (within 72 hours)
* Patients with hepatitis C-positive status may be entered if they have had an intraoperative (back table) biopsy of the transplanted liver or will have a biopsy at the time of randomization. This is not required for patients negative for hepatitis C.

Exclusion Criteria:

* Liver allograft from a living donor or a split liver
* Multiple organ transplant
* Dialysis therapy for >14 days from transplantation to randomization
* History of malignancy in the last 5 years (except hepatoma or non-melanoma skin cancer)
* Previous sirolimus therapy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2005-08; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (34):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - La Jolla, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - Jacksonville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - Newark, New Jersey
  - Hawthorne, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Madison, Wisconsin
- Canada (4):
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - London, Ontario
  - Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 43 study centers in the US and Canada over a period of 3 years (24-Aug-05 to 03-Jul-08)
Pre-assignment Details: Eligible for the study were adult patients (18 to 74 years) who had received a single primary orthotopic liver transplant and were receiving or were scheduled to receive treatment with CellCept® + calcineurin inhibitor (CNI)
Groups:
- CellCept + CNI (Tacrolimus or Cyclosporine): CellCept 1-1.5 g orally or intravenously twice daily, plus a calcineurin inhibitor (CNI) tacrolimus or cyclosporine for 12 months
- CellCept + Sirolimus: CellCept 1-1.5 g orally or intravenously twice daily, plus sirolimus 2-4 mg orally once daily for 9-11 months
Period: Overall Study
Arm/Group | CellCept + CNI (Tacrolimus or Cyclosporine) | CellCept + Sirolimus
Started | 145 | 148
Completed | 96 | 82
Not Completed | 49 | 66

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CellCept + CNI (Tacrolimus or Cyclosporine) | CellCept + Sirolimus | Total
Number analyzed (Participants) | 145 | 148 | 293
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (7.88) | 53.2 (8.83) | 53.3 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 110 | 110 | 220
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 3 | 4 | 7
  Asian or Pacific Islander | 3 | 11 | 14
  Black | 11 | 8 | 19
  White | 126 | 125 | 251
  Other | 2 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] | 173.6 (10.04) | 173.0 (10.26) | 173.3 (10.14)
Weight [Mean (Standard Deviation); unit: kg] | 79 (16.32) | 77.9 (17.56) | 78.4 (16.94)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR) at 12 Months Posttransplant
Description: Mean percent change from baseline in estimated glomerular filtration rate (GFR) calculated by modification of diet in renal disease (MDRD)-6 variable equation at 12 months posttransplantation. MDRD-6 variables: serum creatinine, albumin and urea nitrogen, gender, age and ethnicity.
Time Frame: 12 months posttransplant
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: Percent change in GFR (mL/min)
Arm/Group | CellCept + CNI (Tacrolimus or Cyclosporine) | CellCept + Sirolimus
Number analyzed (Participants) | 124 | 130
Percent change in GFR (mL/min) | 1.2 (39.86) | 19.7 (40.64)
Statistical Analysis 1: Comparison: CellCept + CNI (Tacrolimus or Cyclosporine) vs CellCept + Sirolimus; Test type: Superiority or Other; p = 0.0012, ANCOVA; Mean Difference (Final Values) = 24.9, 95% CI [14.8 to 35.0]

2. Secondary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR) at 6 Months Posttransplant
Description: Mean percent change from baseline in estimated GFR calculated by modification of diet in renal disease (MDRD)-6 variable equation at 6 and 24 months posttransplantation. MDRD-6 variables: serum creatinine, albumin and urea nitrogen, gender, age and ethnicity.
Time Frame: 6 months posttransplant
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: Percent change in GFR (mL/min)
Arm/Group | CellCept + CNI (Tacrolimus or Cyclosporine) | CellCept + Sirolimus
Number analyzed (Participants) | 145 | 148
Percent change in GFR (mL/min) | 1.1 (24.39) | 25.5 (45.82)
Statistical Analysis 1: Comparison: CellCept + CNI (Tacrolimus or Cyclosporine) vs CellCept + Sirolimus; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 25.6, 95% CI [15.7 to 35.6]

3. Secondary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR) at 24 Months Posttransplant
Description: as for outcome 2
Time Frame: 24 months posttransplant
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: Mean percent change in GFR (mL/min)
Arm/Group | CellCept + CNI (Tacrolimus or Cyclosporine) | CellCept + Sirolimus
Number analyzed (Participants) | 124 | 130
Mean percent change in GFR (mL/min) | -8.6 (43.37) | 13.5 (49.17)
Statistical Analysis 1: Comparison: CellCept + CNI (Tacrolimus or Cyclosporine) vs CellCept + Sirolimus; Test type: Superiority or Other; p = 0.0053, ANCOVA; Mean Difference (Final Values) = 28.7, 95% CI [13.7 to 43.7]

4. Secondary Outcome: Change From Baseline in Creatinine Clearance
Description: Mean percent change from baseline in calculated creatinine clearance (CL) at 6, 12, and 24 months posttransplantation
Time Frame: 6, 12, and 24 months posttransplantation
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: Percent change in creatinine CL (mL/min)
Arm/Group | CellCept + CNI (Tacrolimus or Cyclosporine) | CellCept + Sirolimus
Number analyzed (Participants) | 145 | 148
Percent change in creatinine CL (mL/min)
  6 months | -1.3 (23.71) | 18.5 (39.93)
  12 months | -3.0 (35.86) | 14.0 (35.16)
  24 months | -12.8 (41.64) | 7.9 (44.36)
Statistical Analysis 1: Comparison: CellCept + CNI (Tacrolimus or Cyclosporine) vs CellCept + Sirolimus; Statistical analysis for calculated creatinine clearance at 6 months posttransplant; Test type: Superiority or Other; p < 0.0001, ANCOVA; Median Difference (Final Values) = 21.1, 95% CI [12.5 to 29.6]
Statistical Analysis 2: Comparison: CellCept + CNI (Tacrolimus or Cyclosporine) vs CellCept + Sirolimus; Statistical analysis for calculated creatinine clearance at 12 months posttransplant; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 18.2, 95% CI [9.9 to 26.6]
Statistical Analysis 3: Comparison: CellCept + CNI (Tacrolimus or Cyclosporine) vs CellCept + Sirolimus; Statistical analysis for calculated creatinine clearance at 24 months posttransplant; Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = 23.6, 95% CI [10.2 to 37.0]

ADVERSE EVENTS:
Arm/Group | CellCept + CNI (Tacrolimus or Cyclosporine) | CellCept + Sirolimus
Serious Adverse Events (participants affected / at risk) | 65/146 | 67/148
Other Adverse Events (participants affected / at risk) | 134/146 | 141/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CellCept + CNI (Tacrolimus or Cyclosporine) (N=146) | CellCept + Sirolimus (N=148)
Hepatitis C (Infections and infestations) | 10 | 8
Pneumonia (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 3 | 2
Clostridium Difficile Colitis (Infections and infestations) | 1 | 3
Viral Infection (Infections and infestations) | 1 | 1
Abdominal Wall Infection (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridial Infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lactobacillus Infection (Infections and infestations) | 1 | 0
Liver Abscess (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 0
Pseudomonal Sepsis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 2
Peritonitis (Gastrointestinal disorders) | 1 | 1
Umbilical Hernia (Gastrointestinal disorders) | 1 | 1
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 1 | 0
Duodenitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 4 | 4
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 0 | 2
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1
Biliary Anastomosis Complication (Injury, poisoning and procedural complications) | 1 | 0
Complications of Transplanted Kidney (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft Loss (Injury, poisoning and procedural complications) | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 4
Bile Duct Obstruction (Hepatobiliary disorders) | 2 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 1 | 1
Biliary Tract Disorder (Hepatobiliary disorders) | 1 | 1
Hepatic Artery Thrombosis (Hepatobiliary disorders) | 0 | 2
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Haemobilia (Hepatobiliary disorders) | 0 | 1
Hepatic Artery Stenosis (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic Infarction (Hepatobiliary disorders) | 0 | 1
Hepatitis Acute (Hepatobiliary disorders) | 0 | 1
Perforation Bile Duct (Hepatobiliary disorders) | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 7
Chest Pain (General disorders) | 1 | 1
Multi-Organ Failure (General disorders) | 1 | 1
Fat Tissue Increased (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Hernia Obstructive (General disorders) | 0 | 1
Impaired Healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Ulcer Haemorrhage (General disorders) | 0 | 1
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Desmoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epstein-Barr Virus Associated Lymphoproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 4
Embolism Venous (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Neuralgic Amyotrophy (Nervous system disorders) | 0 | 1
Neuroleptic Malignant Syndrome (Nervous system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 5 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0
Liver Function Test Abnormal (Investigations) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Transplant Rejection (Immune system disorders) | 1 | 1
Graft Versus Host Disease (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Liver Transplant Rejection (Immune system disorders) | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Alcohol Abuse (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CellCept + CNI (Tacrolimus or Cyclosporine) (N=146) | CellCept + Sirolimus (N=148)
Diarrhoea (Gastrointestinal disorders) | 42 | 37
Abdominal Pain (Gastrointestinal disorders) | 26 | 21
Nausea (Gastrointestinal disorders) | 23 | 19
Vomiting (Gastrointestinal disorders) | 20 | 12
Abdominal Pain Upper (Gastrointestinal disorders) | 11 | 7
Constipation (Gastrointestinal disorders) | 10 | 6
Mouth Ulceration (Gastrointestinal disorders) | 0 | 10
Stomatitis (Gastrointestinal disorders) | 1 | 9
Hepatitis C (Infections and infestations) | 23 | 20
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 7
Sinusitis (Infections and infestations) | 10 | 4
Nasopharyngitis (Infections and infestations) | 7 | 5
Pyrexia (General disorders) | 21 | 25
Fatigue (General disorders) | 23 | 26
Oedema Peripheral (General disorders) | 17 | 27
Asthenia (General disorders) | 7 | 8
Headache (Nervous system disorders) | 24 | 38
Tremor (Nervous system disorders) | 15 | 12
Dizziness (Nervous system disorders) | 11 | 8
Rash (Skin and subcutaneous tissue disorders) | 5 | 26
Pruritis (Skin and subcutaneous tissue disorders) | 13 | 8
Night Sweats (Skin and subcutaneous tissue disorders) | 6 | 11
Acne (Skin and subcutaneous tissue disorders) | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 11
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 12 | 9
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Hepatic Enzyme Increased (Investigations) | 11 | 12
Liver Function Test Abnormal (Investigations) | 9 | 12
Weight Increased (Investigations) | 8 | 9
Weight Decreased (Investigations) | 10 | 5
White Blood Cell Count Decreased (Investigations) | 9 | 5
Blood Creatinine Increased (Investigations) | 9 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 15
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 2
Anorexia (Metabolism and nutrition disorders) | 6 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 10
Decreased Appetite (Metabolism and nutrition disorders) | 8 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 7
Leukopenia (Blood and lymphatic system disorders) | 21 | 35
Anaemia (Blood and lymphatic system disorders) | 14 | 13
Neutropenia (Blood and lymphatic system disorders) | 11 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Incisional Hernia (Injury, poisoning and procedural complications) | 3 | 9
Incision Site Pain (Injury, poisoning and procedural complications) | 7 | 8
Insomnia (Psychiatric disorders) | 16 | 13
Depression (Psychiatric disorders) | 8 | 10
Hypertension (Vascular disorders) | 15 | 16
Renal Failure (Renal and urinary disorders) | 7 | 2
Jaundice (Hepatobiliary disorders) | 7 | 2

LIMITATIONS AND CAVEATS:
There were no overall limitations and caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.